CLINICAL TRIAL: NCT03813914
Title: Corosolic Acid and Cinnamon for the Treatment of the "Metabolic Syndrome" in Menopausal Transition Women
Brief Title: A New Supplement for the "Metabolic Syndrome"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, Principal Investigator, Clinical professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sineos-3
Record Dates: First submitted 2018-08-07; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
Keywords: insulin resistance, blood pressure,
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sineos (Experimental): Glycyrrhizic acid 38 mg + Cinnamomum Zeylanicum 150 mg + corosolic acid 480 mcg 2 pills/day for 3 months
  Interventions: Dietary Supplement: Sineos
- Placebo comparator (Placebo Comparator): placebo 2 pills/day for 3 months
  Interventions: Dietary Supplement: Sineos

INTERVENTIONS:
Dietary Supplement: Sineos — glycyrrhizic acid 38 mg + Cinnamomum Zeylanicum 150 mg + corosolic acid 480 mcg 2 pills per day

SUMMARY:
This study evaluates the effect of a combination of glycirrhizic acid, Cinnamomun Zeylanicum and corosolic acid for the treatment of metabolic syndrome. Participants receive the supplement or a placebo.

DETAILED DESCRIPTION:
The supplement is composed by of a combination of glycirrhizic acid, Cinnamomun Zeylanicum and corosolic acid. They act in different way reducing insulin resistance, which is the main cause of metabolic syndrome. It was a randomized, controlled study involving 60 women with the metabolic syndrome following the criteria proposed by ATP III in 2015. Main outcomes were the improvement of the parameters that characterizes the metabolic syndrome, such as glucose and insulin levels, triglycerides, HDL-cholesterol and blood pressure.

ELIGIBILITY:
Inclusion Criteria: Postmenopausal women affected by Metabolic Syndrome, diagnosed by ATP 2015 criteria.

-

Exclusion Criteria: treatment with steroids or with hypoglycemic or anti-cholesterol drugs

-

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in glycemia | 3 months
  Reduction of glycemia (mg/dl)
Changes in HDL-cholesterol | 3 months
  Increase of HDL-C (mg/dl)

SECONDARY OUTCOMES:
changes in HOMA-IR | 3 months
  measured as the ratio between glycaemia (mg/dl) and insulin (UI)
changes in total-cholesterol | 3 months
  reduction of cholesterol (mg/dl)
changes in triglycerides | 3 months
  reduction in triglycerides (mg/dl)

IPD SHARING:
Plan to Share IPD: No